CLINICAL TRIAL: NCT00373282
Title: Triamcinolone Acetonide in Silicone-Filled Eyes as Adjunctive Treatment for Proliferative Vitreoretinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8116
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-08

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: PVR; Retinal detachment; Silicone oil; Triamcinolone
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone acetonide

SUMMARY:
To evaluate the effect of triamcinolone acetonide in silicone-filled eyes on the outcome of surgery for PVR.

ELIGIBILITY:
Inclusion Criteria:

* Cases of rhegmatogenous retinal detachment complicated by PVR grade C undergoing vitrectomy and silicone oil tamponade.

Exclusion Criteria:

* History of trauma
* Presence of diabetic retinopathy
* History of vein occlusion
* Giant retinal tear

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Study Completion 2003-06

PRIMARY OUTCOMES:
Single-operation retinal reattachment rate six
months after surgery.

SECONDARY OUTCOMES:
Visual acuity
Retinal reproliferation
Intraocular pressure
Early silicone oil emulsification

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh,MD, Tehran, Tehran Province, Iran